CLINICAL TRIAL: NCT02317237
Title: Anaesthetic Strategy During Endovascular Therapy: General Anaesthesia or Conscious Sedation ?
Brief Title: "GOLIATH" - General Or Local Anaestesia in Intra Arterial THerapy
Acronym: GOLIATH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GOLIATH
Record Dates: First submitted 2014-12-04; First posted 2014-12-15 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2015-11

CONDITIONS: Stroke; Anesthesia; Cerebral Revascularization
MeSH Terms: conditions — Stroke | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Anesthesia (No Intervention): The patients, who will receive general anesthesia during intervention
- Local Anesthesia (Experimental): The patients, who will receive local anesthesia/conscious sedation during intervention
  Interventions: Procedure: Local anesthesia

INTERVENTIONS:
Procedure: Local anesthesia — Conscious sedation
  Arms: Local Anesthesia

SUMMARY:
Patients suffering a stroke with a large vessel occlusion is often treated intra veneous thrombolyse and on top of that also intra arterial therapy. It is unknown what form of anaestesia is best during intra arterial therapy. The investigators will randomize these patients between general anaestesia and local anaestesia. Outcome will be growth of the ischemic lesion as judged on an MRI scan.

ELIGIBILITY:
Inclusion Criteria:

* NIHSS>10
* mRS=<2
* groin puncture<6hours from stroke onset
* occlusion of ICA, ICA-T, M1, M2

Exclusion Criteria:

* MRI contraindications
* GCS<9
* intubated prior to arrival
* posterior circulation stroke
* allergy to anestetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-03-08 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Growth of DWI lesion | 48-72 hours

SECONDARY OUTCOMES:
Time from arrival to groin puncture and recanalization | 1-2 hours
Blood pressure during intervention | 1-2 hours
Modified Rankin Score | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Brekenfeld C, Mattle HP, Schroth G. General is better than local anesthesia during endovascular procedures. Stroke. 2010 Nov;41(11):2716-7. doi: 10.1161/STROKEAHA.110.594622. Epub 2010 Oct 7. No abstract available. PMID 20930156
- [Background] Gupta R. Local is better than general anesthesia during endovascular acute stroke interventions. Stroke. 2010 Nov;41(11):2718-9. doi: 10.1161/STROKEAHA.110.596015. Epub 2010 Oct 7. No abstract available. PMID 20930153
- [Background] Froehler MT, Fifi JT, Majid A, Bhatt A, Ouyang M, McDonagh DL. Anesthesia for endovascular treatment of acute ischemic stroke. Neurology. 2012 Sep 25;79(13 Suppl 1):S167-73. doi: 10.1212/WNL.0b013e31826959c2. PMID 23008394
- [Background] Abou-Chebl A, Lin R, Hussain MS, Jovin TG, Levy EI, Liebeskind DS, Yoo AJ, Hsu DP, Rymer MM, Tayal AH, Zaidat OO, Natarajan SK, Nogueira RG, Nanda A, Tian M, Hao Q, Kalia JS, Nguyen TN, Chen M, Gupta R. Conscious sedation versus general anesthesia during endovascular therapy for acute anterior circulation stroke: preliminary results from a retrospective, multicenter study. Stroke. 2010 Jun;41(6):1175-9. doi: 10.1161/STROKEAHA.109.574129. Epub 2010 Apr 15. PMID 20395617
- [Derived] Tosello R, Riera R, Tosello G, Clezar CN, Amorim JE, Vasconcelos V, Joao BB, Flumignan RL. Type of anaesthesia for acute ischaemic stroke endovascular treatment. Cochrane Database Syst Rev. 2022 Jul 20;7(7):CD013690. doi: 10.1002/14651858.CD013690.pub2. PMID 35857365
- [Derived] Sorensen LH, Speiser L, Karabegovic S, Yoo AJ, Rasmussen M, Sorensen KE, Simonsen CZ. Safety and quality of endovascular therapy under general anesthesia and conscious sedation are comparable: results from the GOLIATH trial. J Neurointerv Surg. 2019 Nov;11(11):1070-1072. doi: 10.1136/neurintsurg-2019-014712. Epub 2019 Mar 29. PMID 30926686
- [Derived] Rasmussen M, Espelund US, Juul N, Yoo AJ, Sorensen LH, Sorensen KE, Johnsen SP, Andersen G, Simonsen CZ. The influence of blood pressure management on neurological outcome in endovascular therapy for acute ischaemic stroke. Br J Anaesth. 2018 Jun;120(6):1287-1294. doi: 10.1016/j.bja.2018.01.039. Epub 2018 Mar 28. PMID 29793595
- [Derived] Simonsen CZ, Yoo AJ, Rasmussen M, Sorensen KE, Leslie-Mazwi T, Andersen G, Sorensen LH. Magnetic Resonance Imaging Selection for Endovascular Stroke Therapy: Workflow in the GOLIATH Trial. Stroke. 2018 Jun;49(6):1402-1406. doi: 10.1161/STROKEAHA.118.021038. Epub 2018 May 8. PMID 29739917
- [Derived] Simonsen CZ, Yoo AJ, Sorensen LH, Juul N, Johnsen SP, Andersen G, Rasmussen M. Effect of General Anesthesia and Conscious Sedation During Endovascular Therapy on Infarct Growth and Clinical Outcomes in Acute Ischemic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2018 Apr 1;75(4):470-477. doi: 10.1001/jamaneurol.2017.4474. PMID 29340574